CLINICAL TRIAL: NCT04193579
Title: Listening to Mom in the Neonatal Intensive Care Unit (NICU): Neural, Clinical and Language Outcomes
Brief Title: Listening to Mom 2: Neural, Clinical and Language Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Katherine E Travis, PhD, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 32638-2; 1K99HD084749-01A1 (NIH); R00HD084749 (NIH)
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Premature Birth
Keywords: Premature Birth; Obstetric Labor, Premature; Obstetric Labor Complications; Pregnancy Complications
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Obstetric Labor Complications; Pregnancy Complications | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Language Treatment Arm (Experimental): An infant participant randomized to the language treatment arm will be played recordings of his/her mother's voice 2-3 hours daily in the intermediate care nursery until discharge.
  Interventions: Behavioral: Language Treatment
- Control Treatment Arm (Sham Comparator): An infant participant randomized to the control treatment arm will receive standard of care. Standard of care does not include being played recordings of his/her mother's voice while admitted to the intermediate care nursery. However, an infant randomized to the control treatment will have the same auditory equipment placed in his/her isolette or crib as an infant randomized to the Language Treatment Arm.
  Interventions: Behavioral: Control Treatment

INTERVENTIONS:
Behavioral: Language Treatment — Recording of a mother's voice reading a children's storybook.
  Arms: Language Treatment Arm
Behavioral: Control Treatment — Standard of Care
  Other Names: Standard of Care
  Arms: Control Treatment Arm

SUMMARY:
The purpose of this study is to examine whether playing recordings of a mother's voice to her infant while in the hospital nursery is an effective treatment for promoting healthy brain and language development in infants born preterm.

DETAILED DESCRIPTION:
Children born preterm are at-risk for developmental language delays. Language problems in preterm children are thought to be related to neurobiological factors, including injuries to white matter structures of the brain and environmental factors, including decreased exposure to maternal speech in the hospital nursery. There is evidence to suggest that maternal speech input may be important for promoting healthy brain and language development.

Participants will be randomly assigned to one of two study groups. Each infant has a 50% chance of being assigned to the group that will listen to a recording of his/her mother's voice and a 50% chance of being assigned to the group that will not be played a voice recording. Mother's of participating infants will have her voice recorded as she reads a common children's storybook. Recordings will be played to infants each day until s/he is discharged from the hospital. To assess the long term impacts of this treatment, research participants and their families will be asked to return for follow-up visiting to perform an MRI brain scan and complete questionnaires and test that assess language development. Follow-up visit occur when infants are between 12 to 18 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Infants born preterm at Stanford Children's Hospital between 24 0/7 - 31 6/7 weeks gestational age

Exclusion Criteria:

* Congenital anomalies
* Recognizable malformation syndromes
* Active seizure disorders
* History of Central Nervous System infections
* Hydrocephalus
* Major sensori-neural hearing loss
* Likelihood to be transferred from NICU to alternate care facility or home environment prior to 36 weeks PMA and/or brain MRI scan
* Intraventricular Hemorrhage Grades III-IV
* Cystic periventricular leukomalacia (PVL)
* Surgical treatment for necrotizing enterocolitis
* Small for gestational age (SGA) <3 percentile and/or Intra-uterine growth restriction (IUGR) no head sparing
* Twin-to-twin transfusions

Ages: 24 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Standard and Raw Scores of Receptive and Expressive Language on MacArthur-Bates Communicative Development Inventory (CDI): Words and Sentences | 18 month follow-up adjusted age for preterm birth
  Parent questionnaire of receptive and expressive language skills. Will be used to assess the long-term impact of intervention on language outcomes. Standard scores are based on percentiles for age and sex and range from <1 to 99th percentile. Raw scores range from 0 to 680. Both higher standard scores and raw scores indicate better performance.

SECONDARY OUTCOMES:
White matter mean diffusivity | Assessed at near-term equivalent age MRI scan (approx. 36-37 weeks postmenstrual age) or at time of hospital discharge, whichever comes first
  Diffusion MRI metric that measures the average rate of water diffusion. It is used to assess white matter development and structure.
Fractional Anisotropy of white matter tracts of the brain | Assessed at near-term equivalent age MRI scan (approx. 36-37 weeks postmenstrual age) or at time of hospital discharge, whichever comes first
  Diffusion MRI metric that measures the directionality of water diffusion in the brain. It is used to assess white matter development and structure.
White matter mean diffusivity | Assessed at 12 month follow-up MRI
  Diffusion MRI metric that measures the average rate of water diffusion. It is used to assess white matter development and structure
Fractional Anisotropy of white matter tracts of the brain | Assessed at 12 month follow-up MRI
  Diffusion MRI metric that measures the directionality of water diffusion in the brain. It is used to assess white matter development and structure.
Score on MacArthur-Bates Communicative Development Inventories: Words and Gestures | 12 month follow-up adjusted for preterm birth
  Parent questionnaire of receptive and expressive language skills. Will be used to assess the long-term impact of intervention on language outcomes. Standard scores are based on percentiles for age and sex and range from <1 to 99th percentile. Raw scores range from 0 to 396. Both higher standard scores and raw scores indicate better performance.
Number of significant apnea, bradycardia and desaturation events requiring stimulation | measured daily and beginning at start of treatment and until end of treatment, approximately 37-40 weeks PMA
  Reflects degree of cardiorespiratory stability
Time (days) to full oral feed | measured daily and beginning at start of treatment and until end of treatment, approximately 37-40 weeks PMA
  days until 100 % of nutrition administered orally
Average daily weight gain | measured daily and beginning at start of treatment and until end of treatment, approximately 37-40 weeks PMA
  measured as weight gain per day

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Travis, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University - Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brignoni-Perez E, Morales MC, Marchman VA, Scala M, Feldman HM, Yeom K, Travis KE. Listening to Mom in the NICU: effects of increased maternal speech exposure on language outcomes and white matter development in infants born very preterm. Trials. 2021 Jul 13;22(1):444. doi: 10.1186/s13063-021-05385-4. PMID 34256820